CLINICAL TRIAL: NCT04822194
Title: Neural Mechanisms of Enhancing Emotion Regulation in Bereaved Spouses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bryan Denny (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor-Investigator, Bryan Denny, Assistant Professor, William Marsh Rice University
Organization: William Marsh Rice University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB-FY2017-90; 1R21AG061597-01A1 (NIH)
Record Dates: First submitted 2021-03-25; First posted 2021-03-30 (Actual); Results first posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Affect; Bereavement; Emotions; Depressive Symptoms; Grief
Keywords: emotion regulation; bereavement; affective neuroscience; social cognitive neuroscience
MeSH Terms: conditions — Depression; Emotional Regulation

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either the "Distancing" or "Reinterpretation" group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Distancing (Experimental): Participants will receive structured cognitive emotion regulation training from an experimenter during an approximately 10-minute interaction in which detailed instructions for implementation of the distancing strategy is explained (i.e. appraising an emotional stimulus as an objective, impartial observer).
  Interventions: Behavioral: Cognitive Emotion Regulation Training
- Reinterpretation (Active Comparator): Participants will receive structured cognitive emotion regulation training from an experimenter during an approximately 10-minute interaction in which detailed instructions for implementation of the reinterpretation strategy is explained (i.e. imagining a better outcome than what initially seemed apparent).
  Interventions: Behavioral: Cognitive Emotion Regulation Training

INTERVENTIONS:
Behavioral: Cognitive Emotion Regulation Training — Cognitive emotion regulation training via cognitive reappraisal involves the ability to modify the trajectory of an emotional response by thinking about and appraising emotional information in an alternative, more adaptive way. Reappraisal to down-regulate negative emotion can be operationalized via two tactics: psychological distancing and reinterpretation. The current study will randomly assign participants to receive a brief course of reappraisal training using either psychological distancing or reinterpretation.

SUMMARY:
This study investigates the underlying mechanisms of a novel emotion regulation intervention among recently bereaved spouses. More specifically, this study examines how thinking about an emotional stimulus in a more adaptive way can affect the relationship between psychological stress, psychophysiological biomarkers of adaptive cardiac response, and brain activity. The emotion regulation strategy targeted is reappraisal, specifically reappraisal-by-distancing (i.e., thinking about a negative situation in a more objective, impartial way) versus reappraisal-by-reinterpretation (i.e., thinking about a better outcome for a negative situation than what initially seemed apparent).

The study seeks to determine if relatively brief, focused reappraisal training in bereaved spouses will result in reduction of self-reported negative affect, increases in respiratory sinus arrhythmia (RSA; a measure of heart rate variability reflecting adaptive cardiac vagal tone), reduction in blood-based inflammatory biomarkers, and changes in neural activity over time. Reappraisal-by-distancing is expected to lead to greater changes in these variables relative to reappraisal-by-reinterpretation. Additionally, it is expected that across time decreases in self-reported negative affect, increases in RSA, reductions in blood-based inflammatory biomarker levels, and changes in neural activity will in turn lead to reductions in depressive symptoms and grief rumination. Finally, it is expected that distancing training will lead to reductions in depressive symptoms and grief rumination that are mediated by changes in the targeted neurobiological and behavioral mechanisms.

DETAILED DESCRIPTION:
The objective of this study is to use an experimental medicine approach to evaluate the basic psychological, psychophysiological, and neural mechanisms underlying a novel cognitive emotion regulation intervention aimed at improving psychological outcomes (e.g., reducing depressive symptoms and grief rumination) in recently bereaved spouses. Cognitive reappraisal (i.e. the ability to modify the trajectory of an emotional response by thinking about and appraising emotional information in an alternative, more adaptive way) represents a highly promising target for psychological intervention in bereavement. Reappraisal can be operationalized via two primary tactics: psychological distancing (i.e. appraising an emotional stimulus as an objective, impartial observer) and reinterpretation (i.e. imagining a better outcome than what initially seemed apparent). The current study builds upon promising preliminary work to investigate the effectiveness and underlying neurobiological mechanisms of a novel, five-session cognitive reappraisal intervention in bereaved spouses.

Recently bereaved participants (i.e. approximately 6 months post-spousal loss) will be randomly assigned to receive training in either distancing or reinterpretation, with five sessions occurring every 1-3 days, with longitudinal collection of affective, psychophysiological, physiological (i.e., blood draws to assess inflammatory biomarkers) and functional magnetic resonance imaging (fMRI) data. Follow-up questionnaire assessments will occur at one- and two-months post-intervention. The study aims to mechanistically relate changes in psychological, psychophysiological, physiological, and neural function during a novel emotion regulation intervention never before implemented in this stressed, high risk group. This research represents a Phase I, Stage I clinical trial. The primary endpoints are the assessments of the psychological, psychophysiological, physiological, and neural mechanisms mediating behavior change as a function of the cognitive emotion regulation intervention. The secondary endpoint is testing the efficacy of the intervention via assessment of psychological outcomes (i.e., the behavior change, as represented in changes in depressive symptoms, stress, and grief rumination).

ELIGIBILITY:
Inclusion Criteria:

* Recent loss of romantic partner within the past 5-7 months
* At least 18 years of age
* Minimum score of 25 on the Inventory for Complicated Grief
* Must be able to speak, read, and write in English
* Must be eligible to safely complete MRI scanning

Exclusion Criteria:

* Death of a second close family member/friend in the past year
* Currently receiving psychotherapy
* Diagnosed with obstructive pulmonary and/or heart disease, diabetes, liver failure, or kidney failure
* Significant visual, auditory, or cognitive impairment
* Divorced within the last year
* Prior participation in a similar emotion regulation training protocol in Dr. Denny's lab
* Any contraindication of MRI scanning (e.g., pregnancy, presence of any non-removable metal on or in the body, implanted medical devices, tattoos, medication patches, orthodontic braces or permanent retainers, hearing aids, history of claustrophobia or breathing disorders)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2024-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Denny, Ph.D., Principal Investigator — William Marsh Rice University
Locations (1):
- Rice University, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Pursuant to the NIH Data Sharing Policy, we have created a Data Sharing Plan for the proposed research. Under this plan, and pursuant to IRB regulations, fully de-identified raw data (defined below) will be made publicly available. Available data will include a compendium of de-identified training condition assignments; raw (i.e. individual subject-by-condition level) negative affect self-reports; questionnaire data; raw heart rate variability data; and raw subject-level brain data (i.e. unpreprocessed functional and structural MRI data, converted to the widely-sharable Brain Imaging Data Structure [BIDS] standard).
Supporting Information: Study Protocol
Time Frame: De-identified data will be made available after the analysis process is complete and research manuscripts are finalized. There is no fixed end date for data access.
Access Criteria: Data will be publicly available on OpenNeuro (https://openneuro.org), a free, open- science neuroinformatics data repository.

REFERENCES:
- [Background] Denny BT, Ochsner KN. Behavioral effects of longitudinal training in cognitive reappraisal. Emotion. 2014 Apr;14(2):425-33. doi: 10.1037/a0035276. Epub 2013 Dec 23. PMID 24364856
- [Background] Denny BT. Getting better over time: A framework for examining the impact of emotion regulation training. Emotion. 2020 Feb;20(1):110-114. doi: 10.1037/emo0000641. PMID 31961188
- [Background] Fagundes CP, Brown RL, Chen MA, Murdock KW, Saucedo L, LeRoy A, Wu EL, Garcini LM, Shahane AD, Baameur F, Heijnen C. Grief, depressive symptoms, and inflammation in the spousally bereaved. Psychoneuroendocrinology. 2019 Feb;100:190-197. doi: 10.1016/j.psyneuen.2018.10.006. Epub 2018 Oct 11. PMID 30368120
- [Background] Bonanno GA, Kaltman S. Toward an integrative perspective on bereavement. Psychol Bull. 1999 Nov;125(6):760-76. doi: 10.1037/0033-2909.125.6.760. PMID 10589301
- [Background] Denny BT, Inhoff MC, Zerubavel N, Davachi L, Ochsner KN. Getting Over It: Long-Lasting Effects of Emotion Regulation on Amygdala Response. Psychol Sci. 2015 Sep;26(9):1377-88. doi: 10.1177/0956797615578863. Epub 2015 Jul 31. PMID 26231911
- [Background] Ochsner KN, Silvers JA, Buhle JT. Functional imaging studies of emotion regulation: a synthetic review and evolving model of the cognitive control of emotion. Ann N Y Acad Sci. 2012 Mar;1251:E1-24. doi: 10.1111/j.1749-6632.2012.06751.x. PMID 23025352
- [Background] Fagundes CP, Murdock KW, LeRoy A, Baameur F, Thayer JF, Heijnen C. Spousal bereavement is associated with more pronounced ex vivo cytokine production and lower heart rate variability: Mechanisms underlying cardiovascular risk? Psychoneuroendocrinology. 2018 Jul;93:65-71. doi: 10.1016/j.psyneuen.2018.04.010. Epub 2018 Apr 13. PMID 29702444

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Distancing | Reinterpretation
Started | 38 | 37
Did Not Receive Emotion Regulation Training | 4 | 0
Discontinued Training | 2 | 4
Lost to Long Term Follow-up | 5 | 7
Completed | 27 (Includes 3 participants that were excluded from analysis (due to incorrect task or scan parameters). Participants that did not complete long-term follow up were still included in analysis if they completed main intervention.) | 26 (Includes 1 participant that was excluded from analysis (due to incorrect task parameters). Participants that did not complete long-term follow up were still included in analysis if they completed main intervention.)
Not Completed | 11 | 11
Not completed — Withdrawal by Subject | 5 | 4
Not completed — Technical issues with MR scanner | 1 | 0
Not completed — Lost to Follow-up | 5 | 7

BASELINE CHARACTERISTICS:
Population: Of the 27 participants to complete distancing protocol, 3 were excluded from analysis due to incorrect task or scan parameters. The 5 lost to follow-up after completion of active intervention were added for a total of 29 distancing participants. Of the 26 participants to complete the reinterpretation protocol, 1 was excluded from analysis due to incorrect task parameters. The 7 lost to follow-up after completion of active intervention were added for a total of 32 reinterpretation participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Distancing | Reinterpretation | Total
Number analyzed (Participants) | 29 | 32 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 11 | 22
  >=65 years | 18 | 21 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.90 (13.48) | 67.22 (9.98) | 67.54 (11.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 21 | 41
  Male | 9 | 11 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 9
  Not Hispanic or Latino | 24 | 25 | 49
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 21 | 28 | 49
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 29 | 32 | 61
Self-reported Negative Affect [Mean (Standard Deviation); unit: units on a scale] — Self-reported negative affect data collected during the emotion regulation task on a 1-4 scale, with 1 meaning "not negative at all" and 4 meaning "very negative".
  units on a scale | 1.98 (0.45) | 2.05 (0.49) | 2.02 (0.46)
Respiratory Sinus Arrhythmia [Mean (Standard Deviation); unit: ln(ms)] — Heart rate variability, or variability in time intervals between heart beats, as measured by the log of root mean square of the successive RR interval differences. RR intervals are interbeat intervals between consecutive heartbeats. Population: Participants that had low quality data (e.g., motion artifacts), recordings that were too short to analyze (less than 150 seconds), or had no recording files available were excluded from analysis.
  ln(ms)
    number analyzed (Participants) | 21 | 24 | 45
    (all) | 3.04 (0.78) | 2.99 (0.78) | 3.01 (0.769)
Neural Activity [Mean (Standard Deviation); unit: units on a scale] — Picture Induced Negative Emotion Signature (PINES) is an independently-defined, validated whole-brain neural pattern map for negative appraisal, with positive weights for areas like the amygdala and insula. PINES Correspondence Scores (PCS) are correlation coefficients derived for each trial type (Look Neutral, Look Negative, Reappraise Negative) per participant by correlating each participant's whole-brain pattern during the task to PINES. PCS correlation coefficients range from -1 to 1, and higher values reflect greater correlation to PINES and thus greater negative affect. Population: Two participants were excluded due to excessive motion artifacts (over 2 mm/degrees).
  units on a scale
    Look Neutral Trials: number analyzed (Participants) | 27 | 32 | 59
    Look Neutral Trials | 0.09 (0.03) | 0.10 (0.03) | 0.10 (0.03)
    Look Negative Trials: number analyzed (Participants) | 27 | 32 | 59
    Look Negative Trials | 0.12 (0.03) | 0.13 (0.03) | 0.13 (0.03)
    Reappraise Negative Trials: number analyzed (Participants) | 27 | 32 | 59
    Reappraise Negative Trials | 0.12 (0.03) | 0.12 (0.04) | 0.12 (0.04)
    Composite Score: number analyzed (Participants) | 27 | 32 | 59
    Composite Score | 0.11 (0.03) | 0.11 (0.04) | 0.11 (0.04)
Grief Rumination [Mean (Standard Deviation); unit: score on a scale] — Grief rumination assessed via Utrecht Grief Rumination Scale (UGRS) and the Inventory for Complicated Grief (ICG). UGRS items are rated from 1 (never) to 5 (very often). Scores range from 15 to 75; higher numbers represent higher grief rumination. These are summed from 3-item subscales Reactions, Injustice, Counterfactuals, Meaning, and Relationships, which all have score ranges of 3-15. Higher scores represent greater grief rumination.
  The ICG assesses grief via 19 first-person statements on a scale of 0 (Never) to 4 (Always) with a range from 0-76. Higher numbers reflect greater grief.
  score on a scale
    Utrecht Grief Rumination Scale (UGRS) Meaning Subscale | 11.17 (2.96) | 12.47 (2.49) | 11.85 (2.78)
    Utrecht Grief Rumination Scale (UGRS) Relationships Subscale | 6.86 (3.37) | 6.00 (3.03) | 6.41 (3.20)
    Utrecht Grief Rumination Scale (UGRS) Counterfactuals Subscale | 7.41 (4.00) | 7.25 (3.55) | 7.33 (3.74)
    Utrecht Grief Rumination Scale (UGRS) Injustice Subscale | 6.79 (3.17) | 6.41 (3.50) | 6.59 (3.32)
    Utrecht Grief Rumination Scale (UGRS) Reactions Subscale | 9.10 (3.00) | 9.22 (2.89) | 9.16 (2.92)
    Utrecht Grief Rumination Scale (UGRS) Composite score | 41.34 (10.54) | 41.34 (11.07) | 41.34 (10.73)
    Inventory for Complicated Grief (ICG) | 27.93 (9.36) | 31.31 (12.10) | 29.70 (10.93)
Depressive Symptoms [Mean (Standard Deviation); unit: score on a scale] — Symptoms of depression assessed via the Center for Epidemiological Studies Depression (CES-D) scale, which asks participants to rate how often in the past week they have experience symptoms of depression, ranging from 0 (Rarely or none of the time) to 3 (Most of the time). Scores range from 0 to 60, with higher scores indicating higher levels of depressive symptoms.
  score on a scale | 26 (8.45) | 23.5 (10.29) | 24.7 (9.47)
Perceived Stress [Mean (Standard Deviation); unit: score on a scale] — Perceived stress assessed via the Perceived Stress Scale (PSS), which consists of 10 self-report items asking participants how often they felt or thought a certain way, ranging from 0 (Never) to 4 (Very Often) with total scores ranging from 0-40. Higher scores indicate higher levels of perceived stress.
  score on a scale | 17.7 (5.74) | 15.9 (7.48) | 16.8 (6.72)

OUTCOME MEASURES:

1. Primary Outcome: Self-reported Negative Affect
Description: Self-reported negative affect data collected during the emotion regulation task on a 1-4 scale, with 1 meaning "not negative at all" and 4 meaning "very negative".
Time Frame: Sessions 1 (baseline/initial session), 2, 3, 4, and 5, which were conducted approximately every 2-3 days over the course of 2 weeks.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Distancing | Reinterpretation
Number analyzed (Participants) | 29 | 32
score on a scale
  Session 2 Negative Affect | 1.88 (0.07) | 1.91 (0.06)
  Session 3 Negative Affect | 1.70 (0.06) | 1.89 (0.06)
  Session 4 Negative Affect | 1.63 (0.06) | 1.85 (0.07)
  Session 5 Negative Affect | 1.63 (0.06) | 1.83 (0.06)
Statistical Analysis 1: Comparison: Distancing vs Reinterpretation; Null hypothesis: no difference between groups. Power analyses using an approximate effect size (d=.70) previously reported for within and between-subjects behavioral analyses of longitudinal reappraisal training data indicate over 95% power (α=.05) to detect within-group effects and 90% power (α=.05) to detect between-group effects require 36 per group; Test type: Superiority; p = 0.053, Mixed Models Analysis; Ran linear mixed model, p-value above reflects group by session interaction

2. Primary Outcome: Respiratory Sinus Arrhythmia
Description: Heart rate variability, or variability in time intervals between heart beats, as measured by the log of the root mean square of the successive RR interval differences (ln(RMSSD)). RR intervals are interbeat intervals between consecutive heartbeats. Average ranges for ln(RMSSD) for 30 to over 75 years of age range from 3.2 to 3.9 for women and 3.2 to 3.8 for men.
Time Frame: as for outcome 1
Population: Participants that had low quality data (e.g., motion artifacts), recordings that were too short to analyze (less than 150 seconds), or had no recording files available were excluded from analysis.
Measure: Mean (Standard Error); unit: ln(ms)
Arm/Group | Distancing | Reinterpretation
Number analyzed (Participants) | 29 | 32
ln(ms)
  Session 2: number analyzed (Participants) | 24 | 27
  Session 2 | 2.80 (0.12) | 2.72 (0.11)
  Session 3: number analyzed (Participants) | 24 | 28
  Session 3 | 2.90 (0.12) | 2.95 (0.14)
  Session 4: number analyzed (Participants) | 24 | 27
  Session 4 | 3.05 (0.15) | 2.84 (0.13)
  Session 5: number analyzed (Participants) | 22 | 28
  Session 5 | 3.09 (0.16) | 2.84 (0.12)
Statistical Analysis 1: Comparison: Distancing vs Reinterpretation; Null hypothesis: no difference between groups. Power analyses using an approximate effect size (d=.70) previously obtained for within and between-subjects analyses of respiratory sinus arrhythmia data indicate over 95% power (α=.05) to detect within-group effects and 90% power (α=.05) to detect between-group effects should be achieved with 36 per group; Test type: Superiority; p = 0.741, Mixed Models Analysis; Ran linear mixed models on natural log of RMSSD, p-value above reflects group by session interaction

3. Primary Outcome: Neural Activity
Description: Picture Induced Negative Emotion Signature (PINES) is an independently-defined, validated whole-brain neural pattern map for negative appraisal, with positive weights for areas like the amygdala and insula. PINES Correspondence Scores (PCS) are correlation coefficients derived for each trial type (Look Neutral, Look Negative, Reappraise Negative) per participant by correlating each participant's whole-brain pattern during the task to PINES. PCS correlation coefficients range from -1 to 1, and higher values reflect greater correlation to PINES and thus greater negative affect.
Time Frame: Sessions 1 (baseline/initial session) and 5, which were conducted approximately 2 weeks apart.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Distancing | Reinterpretation
Number analyzed (Participants) | 27 | 32
units on a scale
  Look Neutral Trials | 0.09 (0.01) | 0.10 (0.005)
  Look Negative Trials | 0.13 (0.01) | 0.14 (0.01)
  Reappraise Negative Trials | 0.11 (0.01) | 0.13 (0.01)
  Composite Score | 0.11 (0.004) | 0.12 (0.003)
Statistical Analysis 1: Comparison: Distancing vs Reinterpretation; Null hypothesis: no difference between groups. Power analyses using a within-subject fMRI effect size estimate for right amygdala affective reactivity from a meta-analysis of Human Connectome Project data of approx. d=.70, applying to between-subjects effects as well, indicate over 95% power (α=.05) to detect within-group effects and 90% power (α=0.05) to detect between-group effects should be achieved with 36 participants per group; Test type: Superiority; p = 0.021, Mixed Models Analysis; Ran linear mixed model, p-value above reflects a group by session interaction

4. Primary Outcome: Grief Rumination
Description: Grief rumination assessed via Utrecht Grief Rumination Scale (UGRS) and the Inventory for Complicated Grief (ICG). UGRS items are rated from 1 (never) to 5 (very often). Scores range from 15 to 75; higher numbers represent higher grief rumination. These are summed from 3-item subscales Reactions, Injustice, Counterfactuals, Meaning, and Relationships, which all have score ranges of 3-15. Higher scores represent greater grief rumination.
  The ICG assesses grief via 19 first-person statements on a scale of 0 (Never) to 4 (Always) with a range from 0-76. Higher numbers reflect greater grief.
Time Frame: Sessions 1 (baseline/initial session) and 5, which were conducted approximately 2 weeks apart, and at the 1- and 2-month follow-ups.
Population: Participants either dropped out or stopped responding during the follow-ups, leading to attrition that lowered our participant number during the 1 and 2 month follow-ups.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Distancing | Reinterpretation
Number analyzed (Participants) | 29 | 32
score on a scale
  Utrecht Grief Rumination Scale Meaning Subscale Session 5 | 10.38 (0.52) | 11.69 (0.51)
  Utrecht Grief Rumination Scale Relationships Subscale Session 5 | 5.66 (0.40) | 5.78 (0.48)
  Utrecht Grief Rumination Scale Counterfactuals Subscale Session 5 | 6.66 (0.66) | 6.81 (0.59)
  Utrecht Grief Rumination Scale Injustice Subscale Session 5 | 5.59 (0.51) | 6.59 (0.66)
  Utrecht Grief Rumination Scale Reactions Subscale Session 5 | 9.24 (0.61) | 9.03 (0.51)
  Utrecht Grief Rumination Scale Composite Score Session 5 | 37.52 (1.85) | 39.91 (2.05)
  Utrecht Grief Rumination Scale Meaning Subscale 1 month follow up: number analyzed (Participants) | 24 | 28
  Utrecht Grief Rumination Scale Meaning Subscale 1 month follow up | 9.42 (0.45) | 10.61 (0.64)
  Utrecht Grief Rumination Scale Relationships Subscale 1 month follow up: number analyzed (Participants) | 24 | 28
  Utrecht Grief Rumination Scale Relationships Subscale 1 month follow up | 6.08 (0.46) | 5.11 (0.34)
  Utrecht Grief Rumination Scale Counterfactuals Subscale 1 month follow up: number analyzed (Participants) | 24 | 28
  Utrecht Grief Rumination Scale Counterfactuals Subscale 1 month follow up | 5.50 (0.52) | 6.11 (0.57)
  Utrecht Grief Rumination Scale Injustice Subscale 1 month follow up: number analyzed (Participants) | 24 | 28
  Utrecht Grief Rumination Scale Injustice Subscale 1 month follow up | 5.13 (0.51) | 5.57 (0.56)
  Utrecht Grief Rumination Scale Reactions Subscale 1 month follow up: number analyzed (Participants) | 24 | 28
  Utrecht Grief Rumination Scale Reactions Subscale 1 month follow up | 8.04 (0.43) | 8.21 (0.55)
  Utrecht Grief Rumination Scale Composite Score 1 month follow up: number analyzed (Participants) | 24 | 28
  Utrecht Grief Rumination Scale Composite Score 1 month follow up | 34.17 (1.56) | 35.61 (1.95)
  Utrecht Grief Rumination Scale Meaning Subscale 2 month follow up: number analyzed (Participants) | 22 | 23
  Utrecht Grief Rumination Scale Meaning Subscale 2 month follow up | 8.77 (0.53) | 10.30 (0.71)
  Utrecht Grief Rumination Scale Relationships Subscale 2 month follow up: number analyzed (Participants) | 22 | 23
  Utrecht Grief Rumination Scale Relationships Subscale 2 month follow up | 5.55 (0.59) | 5.17 (0.55)
  Utrecht Grief Rumination Scale Counterfactuals Subscale 2 month follow up: number analyzed (Participants) | 22 | 23
  Utrecht Grief Rumination Scale Counterfactuals Subscale 2 month follow up | 5.91 (0.69) | 5.48 (0.72)
  Utrecht Grief Rumination Scale Injustice Subscale 2 month follow up: number analyzed (Participants) | 22 | 23
  Utrecht Grief Rumination Scale Injustice Subscale 2 month follow up | 4.05 (0.31) | 5.87 (0.71)
  Utrecht Grief Rumination Scale Reactions Subscale 2 month follow up: number analyzed (Participants) | 22 | 23
  Utrecht Grief Rumination Scale Reactions Subscale 2 month follow up | 6.95 (0.70) | 7.39 (0.75)
  Utrecht Grief Rumination Scale Composite Score 2 month follow up: number analyzed (Participants) | 22 | 23
  Utrecht Grief Rumination Scale Composite Score 2 month follow up | 31.23 (2.24) | 34.22 (2.89)
  Inventory for Complicated Grief Session 5 | 25.41 (1.69) | 29.41 (2.24)
  Inventory for Complicated Grief 1 month follow up: number analyzed (Participants) | 24 | 28
  Inventory for Complicated Grief 1 month follow up | 23.92 (1.77) | 27.32 (2.41)
  Inventory for Complicated Grief 2 month follow up: number analyzed (Participants) | 22 | 23
  Inventory for Complicated Grief 2 month follow up | 21.41 (1.83) | 27.09 (2.55)
Statistical Analysis 1: Comparison: Distancing vs Reinterpretation; Null hypothesis: no difference between groups. Power analyses of an effect size (d=.70) previously reported for within and between-subjects analyses of questionnaire outcomes (i.e., depressive symptoms, grief rumination, perceived stress, reappraisal usage) indicate over 95% power (α=.05) to detect within-group effects and 90% power (α=0.05) for between-group effects should be achieved with 36 per group; Test type: Superiority; p = 0.724, Mixed Models Analysis; We ran linear mixed models, p-value reflects a group by session interaction for the UGRS composite scores
Statistical Analysis 2: Comparison: Distancing vs Reinterpretation; Null hypothesis: no difference between groups; Test type: Superiority; p = 0.835, Mixed Models Analysis; Ran linear mixed model on counterfactuals adjusted for covariates, p-value above reflects group by session interaction
Statistical Analysis 3: Comparison: Distancing vs Reinterpretation; Null hypothesis: no difference between groups; Test type: Superiority; p = 0.090, Mixed Models Analysis; Ran linear mixed model on injustice adjusted for covariates, p-value above reflects group by session interaction
Statistical Analysis 4: Comparison: Distancing vs Reinterpretation; Null hypothesis: no difference between groups; Test type: Superiority; p = 0.983, Mixed Models Analysis; Ran linear mixed model on meaning adjusted for covariates, p-value above reflects group by session interaction
Statistical Analysis 5: Comparison: Distancing vs Reinterpretation; Null hypothesis: no difference between groups; Test type: Superiority; p = 0.760, Mixed Models Analysis; Ran linear mixed model on reaction adjusted for covariates, p-value above reflects group by session interaction
Statistical Analysis 6: Comparison: Distancing vs Reinterpretation; Null hypothesis: no difference between groups; Test type: Superiority; p = 0.402, Mixed Models Analysis; Ran linear mixed model on relations adjusted for covariates, p-value above reflects group by session interaction

5. Primary Outcome: Depressive Symptoms
Description: Symptoms of depression assessed via the Center for Epidemiological Studies Depression (CES-D) scale, which asks participants to rate how often in the past week they have experience symptoms of depression, ranging from 0 (Rarely or none of the time) to 3 (Most of the time). Scores range from 0 to 60, with higher scores indicating higher levels of depressive symptoms.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Distancing | Reinterpretation
Number analyzed (Participants) | 29 | 32
score on a scale
  Center for Epidemiological Studies Depression scale Session 5 | 21.59 (2.04) | 21.78 (1.90)
  Center for Epidemiological Studies Depression scale 1 month follow up: number analyzed (Participants) | 24 | 28
  Center for Epidemiological Studies Depression scale 1 month follow up | 18.96 (1.63) | 20.75 (1.93)
  Center for Epidemiological Studies Depression scale 2 month follow up: number analyzed (Participants) | 22 | 23
  Center for Epidemiological Studies Depression scale 2 month follow up | 16.77 (1.86) | 18.70 (2.07)
Statistical Analysis 1: Comparison: Distancing vs Reinterpretation; Null hypothesis: no difference between groups; Test type: Superiority; p = 0.092, Mixed Models Analysis; We ran a linear mixed model, p-value reflects group by session interaction

6. Primary Outcome: Perceived Stress
Description: Perceived stress assessed via the Perceived Stress Scale (PSS), consisting of 10 self-reported items asking participants how often they felt or thought a certain way, ranging from 0 (Never) to 4 (Very Often). Total range is 0 to 40, with higher scores indicate higher levels of perceived stress.
Time Frame: Sessions 1 (baseline/initial session), 2, 3, 4, and 5, which were conducted approximately every 2-3 days over the course of 2 weeks, and at the 1- and 2- month follow-up.
Population: as for outcome 4
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Distancing | Reinterpretation
Number analyzed (Participants) | 29 | 32
score on a scale
  Perceived Stress Scale Session 2 | 16.07 (1.16) | 15.31 (1.38)
  Perceived Stress Scale Session 3 | 15.93 (1.04) | 15.53 (1.45)
  Perceived Stress Scale Session 4 | 14.52 (1.16) | 14.28 (1.35)
  Perceived Stress Scale Session 5 | 14.41 (1.17) | 14.28 (1.49)
  Perceived Stress Scale 1 month follow up: number analyzed (Participants) | 24 | 28
  Perceived Stress Scale 1 month follow up | 14.29 (1.17) | 14.18 (1.41)
  Perceived Stress Scale 2 month follow up: number analyzed (Participants) | 22 | 23
  Perceived Stress Scale 2 month follow up | 13.00 (1.20) | 12.91 (1.59)
Statistical Analysis 1: Comparison: Distancing vs Reinterpretation; Null hypothesis: no difference between groups; Test type: Superiority; p = 0.585, Mixed Models Analysis; Ran a linear mixed model, p-value reflects group by session interaction

7. Secondary Outcome: Frequency of Reappraisal Usage
Description: Overall reappraisal usage frequency assessed via the Emotion Regulation Questionnaire Reappraisal facet score. Participants report using a 7-point Likert-type scale ranging from 1 (strongly disagree) to 7 (strongly agree). Reappraisal facet scores may range from 6-42. Higher scores represent greater habitual reappraisal usage.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Distancing | Reinterpretation
Number analyzed (Participants) | 29 | 32
score on a scale
  Emotion Regulation Questionnaire Reappraisal facet score Session 1 | 29.86 (1.32) | 30.03 (1.03)
  Emotion Regulation Questionnaire Reappraisal facet score Session 5 | 31.48 (1.08) | 31.69 (0.93)
  Emotion Regulation Questionnaire Reappraisal facet score 1 month follow up: number analyzed (Participants) | 24 | 28
  Emotion Regulation Questionnaire Reappraisal facet score 1 month follow up | 32.17 (1.31) | 31.43 (1.09)
  Emotion Regulation Questionnaire Reappraisal facet score 2 month follow up: number analyzed (Participants) | 22 | 23
  Emotion Regulation Questionnaire Reappraisal facet score 2 month follow up | 31.05 (1.46) | 31.28 (1.35)
Statistical Analysis 1: Comparison: Distancing vs Reinterpretation; Null hypothesis: no difference between groups; Test type: Superiority; p = 0.70, Mixed Models Analysis; Ran linear mixed model, p-value reflects group by session interaction

8. Secondary Outcome: Physical Health
Description: Physical health and quality of life assessed via the RAND 36-Item Short Form Health Survey (SF-36) which assesses 8 subscales: physical functioning, social functioning, role limitations due to physical health problems, body pain, role limitations due to personal or emotional problems, emotional well-being, energy/fatigue, and general health perceptions. Each subscale ranges from 0 to 100, higher scores referring to more adaptive health outcomes.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Distancing | Reinterpretation
Number analyzed (Participants) | 29 | 32
score on a scale
  Physical Function score Session 1: number analyzed (Participants) | 29 | 31
  Physical Function score Session 1 | 77.93 (5.16) | 83.71 (4.21)
  Physical Health score Session 1: number analyzed (Participants) | 29 | 31
  Physical Health score Session 1 | 59.48 (7.17) | 67.74 (6.58)
  Emotional Problems score Session 1: number analyzed (Participants) | 29 | 31
  Emotional Problems score Session 1 | 51.72 (7.51) | 46.24 (7.98)
  Energy score Session 1: number analyzed (Participants) | 29 | 31
  Energy score Session 1 | 48.45 (4.23) | 49.68 (3.67)
  Emotional Wellbeing score Session 1: number analyzed (Participants) | 29 | 31
  Emotional Wellbeing score Session 1 | 62.07 (3.43) | 64.65 (3.37)
  Social Function score Session 1: number analyzed (Participants) | 29 | 31
  Social Function score Session 1 | 68.97 (4.58) | 78.63 (4.61)
  Pain score Session 1: number analyzed (Participants) | 29 | 31
  Pain score Session 1 | 76.47 (4.39) | 71.53 (4.05)
  Health Perceptions score Session 1: number analyzed (Participants) | 29 | 31
  Health Perceptions score Session 1 | 71.55 (4.21) | 71.94 (3.19)
  Physical Function score Session 5 | 80.34 (4.39) | 83.44 (4.14)
  Physical Health score Session 5 | 65.52 (7.59) | 71.09 (5.84)
  Emotional Problems score Session 5 | 57.47 (7.00) | 45.83 (7.14)
  Energy score Session 5 | 49.71 (4.74) | 52.50 (4.07)
  Emotional Wellbeing score Session 5 | 63.17 (3.54) | 64.88 (3.46)
  Social Function score Session 5 | 70.69 (4.49) | 75.39 (4.58)
  Pain score Session 5 | 78.88 (4.02) | 75.70 (4.43)
  Health Perceptions score Session 5 | 71.21 (4.04) | 73.59 (3.49)
  Physical Function score 1 month follow up: number analyzed (Participants) | 24 | 28
  Physical Function score 1 month follow up | 78.75 (4.57) | 85.36 (3.66)
  Physical Health Physical Health score 1 month follow up: number analyzed (Participants) | 24 | 28
  Physical Health Physical Health score 1 month follow up | 62.50 (8.64) | 66.07 (7.84)
  Emotional Problems score 1 month follow up: number analyzed (Participants) | 24 | 28
  Emotional Problems score 1 month follow up | 68.06 (7.89) | 48.81 (7.76)
  Energy score 1 month follow up: number analyzed (Participants) | 24 | 28
  Energy score 1 month follow up | 57.71 (3.91) | 55.54 (3.94)
  Emotional Wellbeing score 1 month follow up: number analyzed (Participants) | 24 | 28
  Emotional Wellbeing score 1 month follow up | 68.17 (2.84) | 68.57 (3.82)
  Social Function score 1 month follow up: number analyzed (Participants) | 24 | 28
  Social Function score 1 month follow up | 81.77 (3.36) | 77.68 (4.56)
  Pain score 1 month follow up: number analyzed (Participants) | 24 | 28
  Pain score 1 month follow up | 75.63 (4.46) | 78.13 (3.97)
  Health Perceptions score 1 month follow up: number analyzed (Participants) | 24 | 28
  Health Perceptions score 1 month follow up | 75.00 (4.13) | 72.32 (3.38)
  Physical Function score 2 month follow up: number analyzed (Participants) | 22 | 23
  Physical Function score 2 month follow up | 79.77 (5.06) | 84.78 (4.75)
  Physical Health score 2 month follow up: number analyzed (Participants) | 22 | 23
  Physical Health score 2 month follow up | 70.45 (8.80) | 66.30 (8.11)
  Emotional Problems score 2 month follow up: number analyzed (Participants) | 22 | 23
  Emotional Problems score 2 month follow up | 80.30 (6.45) | 65.22 (7.97)
  Energy score 2 month follow up: number analyzed (Participants) | 22 | 23
  Energy score 2 month follow up | 55.23 (5.07) | 57.83 (4.47)
  Emotional Wellbeing score 2 month follow up: number analyzed (Participants) | 22 | 23
  Emotional Wellbeing score 2 month follow up | 72.36 (3.36) | 69.74 (3.51)
  Social Function score 2 month follow up: number analyzed (Participants) | 22 | 23
  Social Function score 2 month follow up | 81.82 (4.17) | 80.43 (4.43)
  Pain score 2 month follow up: number analyzed (Participants) | 22 | 23
  Pain score 2 month follow up | 76.70 (4.97) | 76.96 (4.69)
  Health Perceptions Score 2 month follow up: number analyzed (Participants) | 22 | 23
  Health Perceptions Score 2 month follow up | 73.41 (3.93) | 73.04 (4.26)
Statistical Analysis 1: Comparison: Distancing vs Reinterpretation; Null hypothesis: no difference between groups; Test type: Superiority; p = 0.696, Mixed Models Analysis; Ran linear mixed model on emotional problems adjusted for covariates, p-value above reflects group by session interaction
Statistical Analysis 2: Comparison: Distancing vs Reinterpretation; Null hypothesis: no difference between groups; Test type: Superiority; p = 0.452, Mixed Models Analysis; Ran linear mixed model on emotional well-being adjusted for covariates, p-value reflects group by session interaction
Statistical Analysis 3: Comparison: Distancing vs Reinterpretation; Null hypothesis: no difference between groups; Test type: Superiority; p = 0.650, Mixed Models Analysis; Ran a linear mixed model on energy adjusted for covariates, p-value above reflects group by session interaction
Statistical Analysis 4: Comparison: Distancing vs Reinterpretation; Null hypothesis: no difference between groups; Test type: Superiority; p = 0.224, Mixed Models Analysis; Ran linear mixed model on general health perceptions adjusted for covariates, p-value above reflects group by session interaction
Statistical Analysis 5: Comparison: Distancing vs Reinterpretation; Null hypothesis: no difference in groups; Test type: Superiority; p = 0.256, Mixed Models Analysis; Ran linear mixed model on pain adjusted for covariates, p-value above reflects group by session interaction
Statistical Analysis 6: Comparison: Distancing vs Reinterpretation; Null hypothesis: no difference between groups; Test type: Superiority; p = 0.984, Mixed Models Analysis; Ran linear mixed model on physical function adjusted for covariates, p-value above reflects group by session interaction
Statistical Analysis 7: Comparison: Distancing vs Reinterpretation; Null hypothesis: no difference between groups; Test type: Superiority; p = 0.363, Mixed Models Analysis; Ran linear mixed model on physical health adjusted for covariates, p-value above reflects group by session interaction
Statistical Analysis 8: Comparison: Distancing vs Reinterpretation; Null hypothesis: no difference between groups; Test type: Superiority; p = 0.045, Mixed Models Analysis; Ran linear mixed model on social functioning adjusted for covariates, p-value above reflects group by session interaction

9. Secondary Outcome: Inflammatory Biomarkers
Description: Inflammatory biomarkers (e.g., serum IL-6, sIL-6R, IL-10, and TNF- α) measured via blood draw
Time Frame: Sessions 0 and 6, which were conducted approximately 2-3 weeks apart.
Population: Blood biomarkers were a later, secondary addition to the study outcome measures and thus there was not biomarker data collected from each participant. Additionally, attrition from the study accounts for differing participant counts as well.
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Distancing | Reinterpretation
Number analyzed (Participants) | 37 | 31
pg/mL
  IL-10 Session 0: number analyzed (Participants) | 19 | 18
  IL-10 Session 0 | 16.60 (5.19) | 12.60 (4.94)
  Serum IL-6 Session 0: number analyzed (Participants) | 36 | 30
  Serum IL-6 Session 0 | 5.10 (2.24) | 10.34 (3.44)
  TNF- α Session 0: number analyzed (Participants) | 36 | 29
  TNF- α Session 0 | 21.02 (2.27) | 33.53 (5.01)
  sIL-6R Session 0 | 6050.37 (424.24) | 5387.61 (309.64)
  Serum IL-6 Session 6: number analyzed (Participants) | 29 | 27
  Serum IL-6 Session 6 | 5.60 (1.79) | 6.11 (1.63)
  TNF- α Session 6: number analyzed (Participants) | 28 | 26
  TNF- α Session 6 | 23.97 (2.45) | 29.05 (4.24)
  sIL-6R Session 6: number analyzed (Participants) | 30 | 27
  sIL-6R Session 6 | 5931.06 (473.53) | 5494.27 (378.90)
Statistical Analysis 1: Comparison: Distancing vs Reinterpretation; Null hypothesis: no difference between groups; Test type: Superiority; p = 0.422, ANCOVA; Ran a repeated measures ANCOVA of logged IL-6 serum, p-value above reflects time by ER group interaction effect
Statistical Analysis 2: Comparison: Distancing vs Reinterpretation; Null hypothesis: no difference between groups; Test type: Superiority; p = 0.438, ANCOVA; Ran a repeated measures ANCOVA of TNFα, p-value above reflects time by ER group interaction effect

ADVERSE EVENTS:
Time Frame: 3 months
Description: A Serious Adverse Event is a clinical event occurring subsequent to the administration of an agent or intervention which can be characterized as fatal, life-threatening, permanently disabling, requiring hospitalization, or an overdose.
Arm/Group | Distancing | Reinterpretation
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/37
Other Adverse Events (participants affected / at risk) | 0/38 | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2025-05-21): https://cdn.clinicaltrials.gov/large-docs/94/NCT04822194/Prot_000.pdf
  • Statistical Analysis Plan (2025-05-21): https://cdn.clinicaltrials.gov/large-docs/94/NCT04822194/SAP_001.pdf
  • Informed Consent Form (2023-02-15): https://cdn.clinicaltrials.gov/large-docs/94/NCT04822194/ICF_002.pdf